CLINICAL TRIAL: NCT06578637
Title: Investigation of β-hydroxybutyrate Supplementation as Chemoprevention in Familial Adenomatous Polyposis
Acronym: BHB-FAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 08224
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: FAP; Familial Adenomatous Polyposis
Keywords: FAP; Familial adenomatous polyposis; Chemoprevention; Polyps; BHB; Beta-hydroxybutyrate
MeSH Terms: conditions — Adenomatous Polyposis Coli; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A - 10 grams (Experimental): Study participants will take one 35mL dose of HVMN Ketone-IQ by mouth per day (10 total grams of R-1,3-Butanediol) for 2 weeks
  Interventions: Dietary Supplement: R-1,3-Butanediol (10G-A)
- Part A - 20 grams (Experimental): Study participants will take two 35mL dose of HVMN Ketone-IQ by mouth per day (20 total grams of R-1,3-Butanediol) for 2 weeks
  Interventions: Dietary Supplement: R-1,3-Butanediol (20G-A)
- Part A - 30 grams (Experimental): Study participants will take three 35mL dose of HVMN Ketone-IQ by mouth per day (30 total grams of R-1,3-Butanediol) for 2 weeks
  Interventions: Dietary Supplement: R-1,3-Butanediol (30G-A)
- Part B - 30 grams (Experimental): Study participants will take one 35mL dose of HVMN Ketone-IQ by mouth three times per day (30 total grams of R-1,3-Butanediol) for 12 weeks, with a possible additional 12 week extension
  Interventions: Dietary Supplement: R-1,3-Butanediol (30G-B)

INTERVENTIONS:
Dietary Supplement: R-1,3-Butanediol (10G-A) — Study participants will take one 35mL dose of HVMN Ketone-IQ by mouth per day (10 total grams of R-1,3-Butanediol) for 2 weeks
  Other Names: HVMN Ketone-IQ
  Arms: Part A - 10 grams
Dietary Supplement: R-1,3-Butanediol (20G-A) — Study participants will take two 35mL dose of HVMN Ketone-IQ by mouth per day (20 total grams of R-1,3-Butanediol) for 2 weeks
  Other Names: HVMN Ketone-IQ
  Arms: Part A - 20 grams
Dietary Supplement: R-1,3-Butanediol (30G-A) — Study participants will take three 35mL dose of HVMN Ketone-IQ by mouth per day (30 total grams of R-1,3-Butanediol) for 2 weeks
  Other Names: HVMN Ketone-IQ
  Arms: Part A - 30 grams
Dietary Supplement: R-1,3-Butanediol (30G-B) — Study participants will take one 35mL dose of HVMN Ketone-IQ by mouth three times per day (30 total grams of R-1,3-Butanediol) for 12 weeks, with a possible additional 12 week extension
  Other Names: HVMN Ketone-IQ
  Arms: Part B - 30 grams

SUMMARY:
The aim of this study is to evaluate the potential of BHB supplementation as a novel strategy to impede the development and progression of intestinal adenomas in individuals with FAP, thus potentially reducing the need for frequent upper endoscopies and colonoscopies and preventing the need for risk-reducing surgical intervention.

DETAILED DESCRIPTION:
We plan to undertake both an initial absorption study (Part A) in up to 9 individuals with FAP followed by a longitudinal open-label study (Part B) in up to 20 individuals with FAP, who will receive R-1,3-butanediol (HVMN Ketone-IQ), an orally administered BHB precursor. Participants with FAP in Part A will have a blood sample collected and then take R-1,3-butanediol at one of three different doses for 2 weeks, which will be followed by another blood sample collection. In Part B, participants with FAP will undergo colonoscopy/sigmoidoscopy along with an upper endoscopy and will then receive R-1,3-butanediol. The participants will return at 4 weeks and 8 weeks for a blood draw and at that time will also provide a stool sample, and participants will check their ketone levels at home weekly. After 12 weeks of R-1,3-butanediol consumption, an upper endoscopy and colonoscopy/sigmoidoscopy will be performed, which will be the same as the procedure performed on study entry. At this point participants can be finished with the study, or they may have the option of continuing BHB for another 12 weeks in an extension study, followed by a repeat upper endoscopy and colonoscopy/sigmoidoscopy at 24 weeks.

ELIGIBILITY:
Part A

Inclusion Criteria:

1. Have a diagnosis of FAP with genetic testing demonstrating a pathogenic or likely pathogenic germline variant in APC, must have a clinical FAP phenotype with at least one member of the family who has a pathogenic or likely pathogenic germline variant in APC, or must have a clinical diagnosis of FAP as agreed by two gastrointestinal cancer genetics experts
2. Must have an extensive colonic resection with either a subtotal colectomy with ileorectal anastomosis (STC-IRA) or total proctocolectomy with ileal pouch anal anastomosis (TPC-IPAA)
3. Can provide informed consent

Exclusion Criteria:

1. Subject is pregnant, a prisoner, or is under 18 years of age
2. Prior total proctocolectomy with end ileostomy
3. History of inflammatory bowel disease
4. History of diabetes mellitus and are currently on medical diabetes therapy
5. History of chronic kidney disease with an eGFR < 60 mL/min/1.73m2
6. Cancer diagnosis where the subject is receiving active therapy
7. Use of either a ketogenic diet or intermittent fasting (defined as a fasting period of 16 hours or more per day that is not associated with a medical procedure) during the 4 weeks prior to enrollment

Part B

Inclusion Criteria:

1. Have a diagnosis of FAP with genetic testing demonstrating a pathogenic or likely pathogenic germline variant in APC, must have a clinical FAP phenotype with at least one member of the family who has a pathogenic or likely pathogenic germline variant in APC, or must have a clinical diagnosis of FAP as agreed by two gastrointestinal cancer genetics experts.
2. Willing to undergo a colonoscopy or sigmoidoscopy, which may be part of the patient's routine standard care.
3. Able to have a concurrent upper endoscopy performed with the colonoscopy/sigmoidoscopy. This upper endoscopy may be part of the patient's routine standard care.
4. Have at least two colorectal polyps at enrollment (which can be present anywhere in the colon including the rectal cuff, or in the J-pouch [if applicable]).
5. Can provide informed consent.

Exclusion Criteria:

1. Subject is pregnant, a prisoner, or is under 18 years of age
2. Patient is not able to undergo colonoscopy/sigmoidoscopy or upper endoscopy
3. Prior total proctocolectomy with end ileostomy
4. History of inflammatory bowel disease
5. History of diabetes mellitus and are currently on medical diabetes therapy
6. History of chronic kidney disease with an eGFR < 60 mL/min/1.73m2
7. Cancer diagnosis where the subject is receiving active therapy
8. Use of either a ketogenic diet or intermittent fasting (defined as a fasting period of 16 hours or more per day that is not associated with a medical procedure) during the 4 weeks prior to enrollment
9. Regular use of any FAP-related chemopreventive agent in the 6 weeks prior to enrollment including aspirin (> 81mg daily), NSAIDs, BHB supplementation, or any other medication deemed a chemopreventive agent by the study investigators
10. Any colonic or small intestinal polyp observed endoscopically that is > 1 cm in size and is not removed (excluding ampullary adenomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Determine whether oral BHB supplementation is safe and tolerable in FAP | Through study completion, which will be approximately 3 years
  Assessment of FAP patient tolerance of BHB supplements through monitoring of side effects and/or intolerances and patient compliance. We will monitor the percentage of individuals who continue BHB supplementation for the duration of the study, as well as the compliance with taking the BHB supplement.

SECONDARY OUTCOMES:
Measure whether oral BHB supplementations increases serum BHB levels in FAP | Through study completion, which will be approximately 3 years
  Measure fasting serum BHB levels before, during, and at the end of BHB supplementation to determine if BHB supplementation significantly increases serum BHB levels.
Change in transcription and protein expression in the intestinal mucosa and in intestinal polyps in FAP after oral BHB supplementation | Through study completion, which will be approximately 3 years
  Transcriptional profiling and subsequent validation with protein level determination will be performed in the intestinal mucosa and in intestinal polyps before and after BHB supplementation to determine if BHB supplementation is having measurable transcriptional and protein effects on the intestinal mucosa and on intestinal polyps.
Determine whether oral BHB supplementation in FAP reduces intestinal polyp burden | Through study completion, which will be approximately 3 years
  The polyp burden in the duodenum as well as in the lower GI tract (rectal cuff, rectum, rectal pouch) will be calculated through polyp counting and measurement on endoscopy before and after BHB supplementation to permit comparison of polyp burden before and after BHB supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Bryson W Katona, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dmitrieva-Posocco O, Wong AC, Lundgren P, Golos AM, Descamps HC, Dohnalova L, Cramer Z, Tian Y, Yueh B, Eskiocak O, Egervari G, Lan Y, Liu J, Fan J, Kim J, Madhu B, Schneider KM, Khoziainova S, Andreeva N, Wang Q, Li N, Furth EE, Bailis W, Kelsen JR, Hamilton KE, Kaestner KH, Berger SL, Epstein JA, Jain R, Li M, Beyaz S, Lengner CJ, Katona BW, Grivennikov SI, Thaiss CA, Levy M. beta-Hydroxybutyrate suppresses colorectal cancer. Nature. 2022 May;605(7908):160-165. doi: 10.1038/s41586-022-04649-6. Epub 2022 Apr 27. PMID 35477756